CLINICAL TRIAL: NCT01168609
Title: Usefulness of Left Atrial Distensibility to Assess Left Ventricular Filling Pressure and to Predict Prognosis in Acute Myocardial Infarction
Brief Title: Left Atrial Distensibility and Left Ventricular Filling Pressure in Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: No other funding source in this study (Unknown)
Responsible Party: Jong-Khing Huang, MD, Current Superintendent of Kaohsiung Veterans General Hospital
Other Study IDs: VGHKS97-CT4-17
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2007-12

CONDITIONS: Myocardial Infarction
Keywords: Left atrial distensibility; left ventricular filling pressure; tissue Doppler; prognosis; acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with acute myocardial infarction: Acute myocardial infarction (AMI) was defined using the European Society of Cardiology / American College of Cardiology guidelines. Myocardial infarction was detected by the presence of at least two of the following criteria: chest pain lasting more than 30 minutes, typical electrocardiographic changes, and elevated creatinine kinase-MB fraction. Consecutive patients 18 years of age or older who presented within 12 hours after the onset of symptoms were considered for enrollment. Patients who had ST-segment elevation of 1 mm or more in two or more contiguous leads were classified as ST-segment elevation MI.
  Interventions: Procedure: Primary percutaneous coronary intervention

INTERVENTIONS:
Procedure: Primary percutaneous coronary intervention — Primary percutaneous coronary intervention (PCI) and stenting were performed for just the culprit lesion using standard techniques and bare-metal stents in all patients. Unfractionated heparin was used for 3 days after PCI, except in some cases with contraindications, and the dose of unfractionated heparin was selected to prolong the activated partial thromboplastin time by 2-3 times. The decision to use glycoprotein IIb/IIIa inhibitors was left to the discretion of the treating physician. The measurements of LVFP were performed via a fluid-filled pig-tail catheter placed into the LV after coronary angiography if PCI was not indicated or after primary PCI.

SUMMARY:
Left atrial volume (LAV) provides the significant prognostic information in the general population and patients with heart disease, including acute myocardial infarction, left ventricular dysfunction, mitral regurgitation, cardiomyopathy and atrial fibrillation. Large left atrial volume, which represents chronic diastolic dysfunction, is associated with poor outcome, regardless of systolic function. Thereby, LAV provides a long-term view of whether or not the patient has the disease of diastolic dysfunction, regardless of whatever loading conditions are present at the time of the examination, as the hemoglobin A1C in diabetes. However, whether left atrial (LA) parameters could correlate with LVFP and reflect short-term change in left ventricular filling pressure(LVFP) remains unknown. Only one article of our team confirmed the relationship between LAV and LVFP in patients with severe mitral regurgitation by simultaneous echocardiography-catheterization. The prior report proposed a new parameter, LA distensibility, and disclosed its logarithmic relationship with LVFP. The LA distensibility precisely indicated rapid change in LVFP of patients with acute severe mitral regurgitation, and was even superior to mitral E/Em (early-diastolic mitral inflow velocity divided by early-diastolic mitral annular velocity). As left atrial pressure rises to maintain adequate left ventricular diastolic filling, increased atrial wall tension tends to dilate the chamber and stretch the atrial myocardium. Therefore, the smaller left atrial stretchability, the more pressure left atrium (LA) faces to. The first objective of this study was to test the value of LA distensibility for assessing LVFP, particularly in patients with acute myocardial infarction. The second objective was to assess the prognostic value of LA distensibility.

DETAILED DESCRIPTION:
Study population: Between December 2007 and March 2009, this study enrolled AMI patients who had received cardiac catheterization for potential coronary intervention. AMI was defined using the European Society of Cardiology / American College of Cardiology guidelines. Exclusion criteria were the following: 1) presence of mitral stenosis or prosthetic valve, 2) more than mild severity of aortic/mitral valvular problem, 3) any abnormality of atrial septum (e.g., atrial septal defect or aneurysm), 4) rhythm other than sinus rhythm and 5) lack of informed consent. Finally, 521 patients participated in this study and were under final analysis. All patients and controls gave written informed consent to participate in the study, and the study was approved by the institutional review board at Kaohsiung Veterans General Hospital.

Cardiac catheterization: Before catheterization, all patients received 300 mg of aspirin and 300 mg of clopidogrel. After detail explanation and informed consent, patients were subjected to diagnostic coronary angiography via a femoral approach following intravenous injection of unfractionated 7500 U heparin. There were 46 cases required coronary artery bypass grafting (CABG) with/without other repair procedures due to failed percutaneous coronary intervention procedure, severe multiple vessel disease, left main lesion, cardiac rupture, severe mitral regurgitation or post-MI ventricular septal defect. All other patients were treated successfully by primary PCI and stenting. Eight patients who had initially received primary PCI were later treated by CABG due to failure of the procedure, severe multiple vessel disease or complications (the 46 CABG patients cited above included these eight patients). Coronary angioplasty and stenting were performed for just the culprit lesion using standard techniques and bare-metal stents in all patients. The decision to use glycoprotein IIb/IIIa inhibitors was left to the discretion of the treating physician. The measurements of LVFP were performed via a fluid-filled pig-tail catheter placed into the LV after coronary angiography if PCI was not indicated or after primary PCI. The LVFP was continuously recorded (50 mm/s) by a 6-F pigtail catheter placed at the apex of the left ventricle and was taken from 3 to 5 end-respiratory cycles if patients could tolerate breath holding. The LVFP value was calculated as the mean of at least 3 consecutive cardiac cycles.

Echocardiographic and myocardial tissue Doppler measurements: Echocardiography was performed immediately after LVFP measurements. All studies were performed by experienced sonographers and the results were reviewed by staff cardiologists with advanced echocardiography training. Left ventricular ejection fraction was calculated using Simpson's method for biplane images. Pulsed-wave tissue Doppler imaging (TDI) was performed using spectral pulsed Doppler signal filters, by adjusting the Nyquist limit to 15 - 20 cm/s (which approximated the myocardial velocities) and using the minimum optimal gain. In the apical views, a 3-mm, a pulsed-wave Doppler sample volume was placed at the level of the mitral annulus over the septal, lateral and inferior borders. Pulsed-wave TDI results were characterized by a myocardial systolic wave (Sm) and 2 diastolic waves: early (Em) and atrial contraction (Am). The pulsed-wave TDI tracing was recorded over 5 cardiac cycles at a sweep speed of 100 mm/s and was used for offline calculations. Average Em of septal and lateral mitral annulus was chose to estimate LVFP by the method of mitral E/Em.

Measurement of LA volume: All volume measurements were calculated from apical four- and two-chamber views using the biplane area-length method. The LA volumes were measured at three points: 1) immediately before the mitral valve opening (maximal LV volume or Volmax); 2) at onset of the P-wave on electrocardiography (pre-atrial contraction volume or Volp); and 3) at mitral valve closure (minimal LV volume or Volmin). The LA distensibility was calculated as (Volmax - Volmin) / Volmin. The LA ejection fraction was calculated as (Volp - Volmin) / Volp. In all patients, LA volumes were indexed to body surface area (BSA).

Follow-up: During index hospitalization, only cardiovascular death was deemed an event. A follow-up survey assessing inhospital mortality and hard events was carried out after discharge of index hospitalization. Sudden cardiac death, death related to cardiovascular problem, and any hospitalization related to heart were defined as hard event. Death within 1 hour of the onset of acute illness or sudden collapse with unknown cause was diagnosed as sudden cardiac death. Follow-up was performed between December 2007 and February 2010 by telephone interviews, medical record reviews, and home visits.

Interobserver variability: In the first fifty enrolled cases, Volmax, Volmin, and Volp were measured by two independent observers. Interobserver variability was calculated as the difference between the values obtained by the two observers divided by the mean. Interobserver difference and variability of Volmax were 4.1±5.4 ml and 6.6±8.7%, respectively. Interobserver variabilities and differences, were 8.1±8.9% and 2.9±3.2 ml for Volmin, 6.7±7.4% and 3.1±3.4 for Volp, respectively. Therefore, interobserver variabilities in LA distensibility and LA ejection fraction measurements were 7.8±6.6% and 3.1±3.2%, respectively.

Statistical analysis: The SPSS software was used for all statistical analyses. Baseline characteristics of the study patients were grouped according to quartile of LA distensibility. All continuous variables were presented as means ± standard deviation. Analysis of variance and post hoc test for unpaired data were used to evaluate the significance of differences between groups. A p vale of < 0.05 was considered statistically significant. Comparison of clinical characteristics was performed by chi-square analysis for categorical variables. Event-free survival curves were generated by means of Kaplan-Meier estimates, and differences in survival were compared with use of the log-rank test. To evaluate the effect of different levels of LA distensibility on in-hospital mortality, and hard events, relative risk and 95% confidence intervals were calculated as hazard ratios derived from the Cox proportional-hazards model. Multivariate models were fitted with use of the available clinical covariates. The relationship curve between LA distensibility and LVFP was estimated using SPSS software. Bivariate analysis, simple correlation and linear regression were used when appropriate. Receiver-Operating Characteristic (ROC) curve analysis was also performed to assess the sensitivity and specificity for predicting elevated LVFP (> 15 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction was detected by the presence of at least two of the following criteria: chest pain lasting more than 30 minutes, typical electrocardiographic changes, and elevated creatinine kinase-MB fraction. Consecutive patients 18 years of age or older who presented within 12 hours after the onset of acute myocardial infarction were considered for enrollment.

Exclusion Criteria:

* 1) presence of mitral stenosis or prosthetic mitral valves
* 2) more than mild severity of aortic/mitral valvular problem
* 3) any abnormality of atrial septum (e.g., atrial septal defect or aneurysm)
* 4) rhythm other than sinus rhythm
* 5) inadequate image quality
* 6) lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between December 2007 and March 2009, this study enrolled AMI patients who had received cardiac catheterization for potential percutaneous coronary intervention (PCI). Myocardial infarction was detected by the presence of at least two of the following criteria: chest pain lasting more than 30 minutes, typical electrocardiographic changes, and elevated creatinine kinase-MB fraction. Consecutive patients 18 years of age or older who presented within 12 hours after the onset of symptoms were considered for enrollment. Patients who had ST-segment elevation of 1 mm or more in two or more contiguous leads were classified as ST-segment elevation MI. Others were classified as non ST-segment elevation MI. .
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
in-hospital death after acute myocardial infarction | Average 2 weeks
  All cause mortality during index hospitalization of acute myocardial infarction was recorded.

SECONDARY OUTCOMES:
1-year hard event rate after acute myocardial infarction | 1 year after discharge
  After index hospitalization, patients were followed up at our cardiovascular clinic for at least 1 year. A follow-up survey assessing hard cardiovascular (CV) events was carried out after discharge. All cause mortality and heart failure with re-hospitalization were defined as hard CV event. Follow-up was performed between December 2007 and February 2010 by telephone interviews, medical record reviews, and home visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Khing Huang, MD, Study Chair — Department of Medical Education and Research Kaohsiung Veterans General Hospital
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Taiwan

REFERENCES:
- [Result] Hsiao SH, Huang WC, Lin KL, Chiou KR, Kuo FY, Lin SK, Cheng CC. Left atrial distensibility and left ventricular filling pressure in acute versus chronic severe mitral regurgitation. Am J Cardiol. 2010 Mar 1;105(5):709-15. doi: 10.1016/j.amjcard.2009.10.052. PMID 20185021
- See also: Government Research Bulletin — http://www.grb.gov.tw/index.htm